CLINICAL TRIAL: NCT05422222
Title: A Phase 3 Study Evaluating the Pharmacokinetics, Safety, and Tolerability of VX-121/Tezacaftor/Deutivacaftor Triple Combination Therapy in Cystic Fibrosis Subjects 1 Through 11 Years of Age
Brief Title: Evaluation of VX-121/Tezacaftor/Deutivacaftor in Cystic Fibrosis (CF) Participants 1 Through 11 Years of Age
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VX21-121-105; 2024-513754-29-00 (Other: EU Trial (CTIS) Number)
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: VX-121/TEZ/D-IVA (Experimental): Participants will receive VX-121/TEZ/D-IVA in the morning.
  Interventions: Drug: VX-121/TEZ/D-IVA
- Part B: VX-121/TEZ/D-IVA (Experimental): Participants will receive VX-121/TEZ/D-IVA in the morning with the dose(s) to be based on the outcome of Part A.
  Interventions: Drug: VX-121/TEZ/D-IVA

INTERVENTIONS:
Drug: VX-121/TEZ/D-IVA — Fixed-dose combination for oral administration.
  Other Names: VX-121/VX-661/VX-561; VX-121/VX-661/CTP-656; VX-121/tezacaftor/deutivacaftor

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics, safety, tolerability and efficacy of VX-121/tezacaftor/deutivacaftor (VX-121/TEZ/D-IVA) in CF participants with at least 1 triple combination responsive (TCR) mutation in the cystic fibrosis transmembrane conductance regulator (CFTR) gene.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with stable CF and at least 1 TCR mutation (including F508del) in the CFTR gene

Key Exclusion Criteria:

* History of solid organ, hematological transplantation, or cancer
* Hepatic cirrhosis with portal hypertension, moderate hepatic impairment (Child Pugh Score 7 to 9), or severe hepatic impairment (Child Pugh Score 10 to 15)
* Lung infection with organisms associated with a more rapid decline in pulmonary status

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Part A: Observed Pre-dose Plasma Concentration (Ctrough) of VX-121, TEZ, D-IVA, and Relevant Metabolites | From Day 1 up to Day 22
Part A: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 50
Part B: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Week 28

SECONDARY OUTCOMES:
Part B: Absolute Change in Sweat Chloride (SwCl) | From Baseline Through Week 24
Part B: Observed Pre-dose Plasma Concentration (Ctrough) of VX-121, TEZ, D-IVA, and Relevant Metabolites | From Day 1 up to Week 16
Part B: Drug Acceptability Assessment Using Modified Facial Hedonic Scale | At Day 1 and Week 24
Part B: Absolute Change in Percent Predicted Forced Expiratory Volume (ppFEV1) | From Baseline Through Week 24
Part B: Number of Pulmonary Exacerbation (PEx) | From Baseline Through Week 24
Part B: Number of CF-Related Hospitalizations | From Baseline Through Week 24
Part B: Absolute Change in Cystic Fibrosis Questionnaire-Revised (CFQ-R) Respiratory Domain (RD) Score | From Baseline Through Week 24
Part B: Absolute Change in Body Mass Index (BMI) | From Baseline at Week 24
Part B: Absolute Change in BMI-for-age Z-score | From Baseline at Week 24
Part B: Absolute Change in Weight | From Baseline at Week 24
Part B: Absolute Change in Weight-for-age Z-score | From Baseline at Week 24
Part B: Absolute Change in Weight-for-length | From Baseline at Week 24
Part B: Absolute Change in Weight-for-length Z-score | From Baseline at Week 24
Part B: Absolute Change in Height | From Baseline at Week 24
Part B: Absolute Change in Height-for-age Z-score | From Baseline at Week 24
Part B: Absolute Change in Length | From Baseline at Week 24
Part B: Absolute Change in Length-for-age Z-score | From Baseline at Week 24
Part B: Proportion of Participants With SwCl <60 millimole per liter (mmol/L) | From Baseline Through Week 24
Part B: Proportion of Participants With SwCl <30 mmol/L | From Baseline Through Week 24

CONTACTS AND LOCATIONS:
Locations (38):
- United States (19):
  - Children's Hospital of Orange County, Orange, California
  - Stanford University Clinical and Translational Research Unit, Palo Alto, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - The Emory Clinic / Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children at Indiana University Health, Indianapolis, Indiana
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Respiratory and Critical Care Specialists, P.A., Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Washington University School of Medicine / St. Louis Children's Hospital, St Louis, Missouri
  - Cohen Children's Medical Center, Lake Success, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Children's Hospital/University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital - Wallace Tower, Houston, Texas
  - Vermont Lung Center, Colchester, Vermont
  - American Family Childrens Hospital, Madison, Wisconsin
- Australia (4):
  - The Kids Research Institute Australia, Nedlands
  - Women's and Children's Hospital, North Adelaide
  - The Royal Children's Hospital, Parkville
  - Queensland Children's Hospital, South Brisbane
- Canada (2):
  - The Hospital for Sick Children, Toronto
  - British Columbia Children's Hospital, Vancouver
- France (2):
  - CHU Lyon - Hopital Femme Mere-Enfant, Bron
  - Hopital Necker, Enfants Malades, Paris
- Germany (3):
  - Charité Universitätsmedizin BerlinX, Berlin
  - Kinderklinik III, Abt. fur Pneumologie, Essen
  - Medizinische Hochschule Hannover, Hanover
- Erasmus Medical Center / Sophia Children's Hospital, Rotterdam, Netherlands
- Starship Children's Hospital, Grafton, New Zealand
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Karolinska Universitetssjukhuset, Huddinge, Stockholm
- Switzerland (2):
  - Inselspital - Universitaetsspital Bern, Bern
  - Kinderspital Zurich, Zurich
- United Kingdom (2):
  - Children and Young Adults Research Unit, Cardiff
  - Great Ormond Street Hospital for Children, London

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/

REFERENCES:
- [Derived] Hoppe JE, Kasi AS, Pittman JE, Jensen R, Thia LP, Robinson P, Tirakitsoontorn P, Ramsey B, Mall MA, Taylor-Cousar JL, McKone EF, Tullis E, Salinas DB, Zhu J, Chen YC, Rodriguez-Romero V, Sosnay PR, Davies G; VX21-121-105 Study Group. Vanzacaftor-tezacaftor-deutivacaftor for children aged 6-11 years with cystic fibrosis (RIDGELINE Trial VX21-121-105): an analysis from a single-arm, phase 3 trial. Lancet Respir Med. 2025 Mar;13(3):244-255. doi: 10.1016/S2213-2600(24)00407-7. Epub 2025 Jan 2. PMID 39756425